CLINICAL TRIAL: NCT06904781
Title: Treatment Outcomes of Pulpotomy Versus Pulpectomy in Vital Primary Molars Diagnosed With Symptomatic Irreversible Pulpitis: A Non-inferiority Randomised Controlled Trial
Brief Title: Treatment Outcomes of Pulpotomy Versus Pulpectomy in Vital Primary Molars Diagnosed With Irreversible Pulpitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Jordan University of Science and Technology (Other); Primary Health Care Corporation, Qatar (Other Government); Cairo University (Other); Christian Dental College (Unknown); Oral and Dental Teaching Hospital, Libya (Unknown)
Responsible Party: Principal Investigator, Nebu Philip, Assistant Professor, Qatar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025_RCT
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Irreversible Pulpitis
Keywords: Pulpectomy; Pulpotomy; Vital primary molars; Irreversible pulpitis
MeSH Terms: interventions — Pulpotomy; Pulpectomy

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulpotomy (Experimental): Participants diagnosed with symptomatic irreversible pulpitis in vital primary molars will receive the pulpotomy treatment intervention
  Interventions: Procedure: Pulpotomy
- Pulpectomy (Active Comparator): Participants diagnosed with symptomatic irreversible pulpitis in vital primary molars will receive the pulpectomy treatment intervention.
  Interventions: Procedure: Pulpectomy

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy is a conservative pulp treatment option where only the coronal pulp is removed and a bioactive medicament (MTA) is placed over the remnant radicular pulp after haemostasis is achieved.
  Arms: Pulpotomy
Procedure: Pulpectomy — Pulpectomy is treatment procedure in primary teeth where the entire coronal and radicular pulp is extirpated and the root canal system filled with a resorbable material (Vitapex/Metapex)
  Arms: Pulpectomy

SUMMARY:
This randomised controlled trial aims to compare treatment outcomes between pulpotomy and pulpectomy when used to treat vital primary molars diagnosed with symptomatic irreversible pulpitis. Compared to the standard pulpectomy treatment, pulpotomy is a technically simpler procedure, less time consuming, easier for young patients to tolerate, while retaining the proprioceptive sensation of the tooth - all important advantages when treating young children.

DETAILED DESCRIPTION:
Background: Pulpectomy continues to be the standard treatment recommendation for management of vital primary molars diagnosed with symptomatic irreversible pulpitis. The recent decade has seen a paradigm shift in the treatment concepts of how vital mature permanent molars diagnosed with irreversible pulpitis can be more conservatively managed using vital pulp therapy techniques like pulpotomy. However, despite emerging evidence indicating similarities between primary and permanent tooth pulp response to dental caries, there is limited research on whether pulpotomy can be similarly used as a definitive treatment modality for vital primary teeth with irreversible pulpitis. This randomised controlled trial (RCT) aims to compare the treatment effectiveness of pulpotomy versus pulpectomy in management of vital primary molars diagnosed with symptomatic irreversible pulpitis over a two-year period.

Methods/Design: This clinical study is a parallel, two-armed, open label, non-inferiority RCT with a 1:1 allocation ratio between the experimental intervention arm (pulpotomy) and the active comparator arm (pulpectomy). Healthy cooperative children, between 4-9 years of age, who have painful primary molars with clinical symptoms typical of irreversible pulpitis will be recruited after obtaining informed consent from their parents/legal guardians. 80 vital primary molars clinically diagnosed with symptomatic irreversible pulpitis will be randomly distributed between the two treatment arms. The primary outcomes that will be assessed are clinical success after one-year and two-years of the trial interventions. The influence of baseline pre-operative variables (age; gender; tooth type; site of caries; pre-operative furcal radiolucency; pre-operative pain intensity) and intra-operative factors (time taken to achieve haemostasis) on treatment outcomes will also be assessed. The secondary outcomes evaluated will be the immediate (24 h and 7 d) post-operative pain relief afforded by the two treatment interventions, and the radiographic success after one-year and two-years of the trial interventions.

Discussion: This trial seeks to provide evidence on whether pulpotomy treatment can be no worse than the standard pulpectomy treatment for the management of symptomatic irreversible pulpitis in vital primary molars.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (ASA I and II) co-operative children (Frankl Scale + and ++) between the ages of four and nine years.
2. Participants have symptoms typical of irreversible pulpitis in one of the primary molars.
3. The pulp of the affected primary molar is vital.
4. Radicular pulp health is confirmed by attainment of radicular pulp haemostasis within 6 minutes of coronal pulp amputation.
5. The affected primary molars can be restored with full coverage stainless steel crowns.
6. Any physiologic root resorption, if present, is less than ⅓ the root length.

Exclusion Criteria:

1. Clinical examination of affected primary molar reveals signs of pulpal infection (e.g. pathologic tooth mobility, parulis/fistula, or soft tissue swelling).
2. Pre-operative periapical radiograph suggests presence of periapical radiolucency or pathologic root resorption.
3. Visual examination of pulp tissue after deroofing reveals signs of necrosis (e.g. avascular/minimally bleeding pulp tissue or yellowish necrotic areas/purulent exudate).
4. Signs of extensive radicular pulp inflammation i.e., root pulp bleeding continues even after 6-min.
5. Parents not willing to place full coverage crowns post-treatment.
6. Clinical diagnosis of irreversible pulpitis between two adjacent primary molars is not sharply defined.
7. Unable to perform clinical procedure under rubber dam

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-treatment clinical outcomes based on presence/absence of pain, tenderness, or signs of infection/pathologic mobility | 6 months; 12 months; 24 months
  Clinical outcome success will be determined at 6-, 12-, and 24-months based on the treated tooth meeting all the below criteria: (i) Treated tooth is not associated with any pain or discomfort; (ii) Treated tooth is not associated with tenderness on percussion or palpation; (iii) Treated tooth is not associated with any swelling, parulis, or fistula; (iv) Treated tooth is not associated with any pathological mobility

SECONDARY OUTCOMES:
Post-treatment radiographic outcomes based on presence/absence of pathologic root resorption, new furcal or periapical lesions, or size change of any pre-treatment furcal rarefaction | 6 months; 12 months; 24 months
  Radiographic outcome success will be determined at 6-, 12-, and 24-months based on the pulpotomy treated tooth meeting all the below criteria: - No signs of pathological internal/external root resorption or new furcal/periapical lesions on recall periapical radiographs - Complete radiographic healing or reduction/no change in size of any pre-treatment furcal rarefaction on recall periapical radiographs
Immediate post-treatment pain relief | 24 hours; 7 day
  Pain scores that will be recorded at 24-hours and 7-days post-treatment using a child friendly Visual Analogue Scale (VAS). The VAS has five-point pain score: 0-No Pain; 1-Mild Pain; 2-Moderate Pain; 3-Severe Pain; and 4-Very Severe Pain. This VAS pain score will be used to evaluate pain reduction afforded by the treatment intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nebu Philip, MDS, PhD, Principal Investigator — Qatar University

IPD SHARING:
Plan to Share IPD: No